CLINICAL TRIAL: NCT01864135
Title: Improved Prostate Cancer Diagnosis - Combination of Magnetic Resonance Imaging
Brief Title: Improved Prostate Cancer Diagnosis - Combination of Magnetic Resonance Imaging and Biomarkers
Acronym: IMPROD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: University of Turku (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 112/180/2012
Record Dates: First submitted 2013-04-17; First posted 2013-05-29 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MRI (Experimental): Comparison of targeted transrectal ultrasound guided prostate biopsies based on 3T multiparametric MRI findings to systematic non-targeted transrectal ultrasound guided prostate biopsies
  Interventions: Device: 3T MRI (Magnetom Verio 3T, Erlangen, Germany); Device: Transrectal ultrasound (Bk Medical Pro Focus Ultraview 2202 system)

INTERVENTIONS:
Device: 3T MRI (Magnetom Verio 3T, Erlangen, Germany)
Device: Transrectal ultrasound (Bk Medical Pro Focus Ultraview 2202 system)

SUMMARY:
Prostate cancer has been the most common cancer in men in Finland over the last ten years. Prostate-specific antigen (PSA) plays an important role in screening of prostate cancer. However, PSA has a limited sensitivity and specificity for prostate cancer detection. Commonly, the diagnosis of prostate cancer is done by transrectal ultrasonography (TRUS) guided biopsy. Due to the low accuracy of TRUS, a systematic biopsy is usually performed instead of targeted TRUS biopsy. As biopsy carries a risk of increase in complications, there is an increasing interest in developing more accurate non-invasive imaging modalities.

This study will enroll 150 men with clinical suspicion of prostate cancer due to higher serum level of PSA than 2.5 ng/ml and/or abnormal digital rectal examination. Multiparametric magnetic resonance imaging (mpMRI) at 3 Tesla (T) magnetic field using surface coils will be used to non-invasively predict the presence or absence of prostate cancer. Targeted TRUS guided biopsy based on MRI findings will be performed in addition to routine twelve core TRUS biopsy. Moreover, selected serum and urine biomarkers as well as biomarkers extracted from fresh biopsy sample will be collected and correlated with the presence or absence of prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age: 40 to 85 years
* Clinical suspicion of prostate cancer based on: serum level of PSA from 2,5 ng/ml to 25 ng/ml in two following measurements and/or abnormal digital rectal examination
* Mental status: Patients must be able to understand the meaning of the study
* Informed consent: The patient must sign the appropriate Ethics Committee (EC) approved informed consent documents in the presence of the designated staff

Exclusion Criteria:

* previous prostate biopsy in the last 6 months
* previous diagnosis of prostate carcinoma
* previous prostate surgeries, e.g. TURP (transurethral prostatic resection)
* symptomatic of acute prostatitis
* contraindications for MRI (cardiac pacemaker, intracranial clips etc)
* uncontrolled serious infection
* claustrophobia
* any other conditions that might compromise patients safety, based on the clinical judgment of the responsible urologist

Ages: 40 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2013-03; Primary Completion 2015-02 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of multiparametric MRI in prostate cancer diagnosis | 3 months
  Multiparametric MRI is performed in patients with clinical suspicion of prostate cancer (elevated PSA and/or abnormal DRE). The accuracy will be determined using the results from transrectal ultrasound guided biopsies.

SECONDARY OUTCOMES:
Predictive value of molecular markers to estimate prostate cancer diagnosis. | 3 months
  molecular markers include PCR-analyses of multiple markers from biopsy material. The association of molecular marker status is used to estimate the risk of prostate cancer on biopsies.

CONTACTS AND LOCATIONS:
Overall Officials: Hannu J Aronen, MD, PhD, Principal Investigator — Department of Diagnostic Radiology, University of Turku
Locations (1):
- Turku University Hospital, Turku, Finland

REFERENCES:
- [Derived] Khan MFL, Soikkeli M, Routila E, Krannila S, Terava J, Taimen P, Bostrom PJ, Pettersson K. Clinical Utility of Mutant Antibody-Based Assays for Determination of Internally Cleaved and Intact Forms of Free Prostate-Specific Antigen. J Appl Lab Med. 2019 May;3(6):1014-1021. doi: 10.1373/jalm.2018.027797. Epub 2019 Feb 1. PMID 31639692
- [Derived] Montoya Perez I, Jambor I, Pahikkala T, Airola A, Merisaari H, Saunavaara J, Alinezhad S, Vaananen RM, Tallgren T, Verho J, Kiviniemi A, Ettala O, Knaapila J, Syvanen KT, Kallajoki M, Vainio P, Aronen HJ, Pettersson K, Bostrom PJ, Taimen P. Prostate Cancer Risk Stratification in Men With a Clinical Suspicion of Prostate Cancer Using a Unique Biparametric MRI and Expression of 11 Genes in Apparently Benign Tissue: Evaluation Using Machine-Learning Techniques. J Magn Reson Imaging. 2020 May;51(5):1540-1553. doi: 10.1002/jmri.26945. Epub 2019 Oct 6. PMID 31588660
- [Derived] Jambor I, Verho J, Ettala O, Knaapila J, Taimen P, Syvanen KT, Kiviniemi A, Kahkonen E, Perez IM, Seppanen M, Rannikko A, Oksanen O, Riikonen J, Vimpeli SM, Kauko T, Merisaari H, Kallajoki M, Mirtti T, Lamminen T, Saunavaara J, Aronen HJ, Bostrom PJ. Validation of IMPROD biparametric MRI in men with clinically suspected prostate cancer: A prospective multi-institutional trial. PLoS Med. 2019 Jun 3;16(6):e1002813. doi: 10.1371/journal.pmed.1002813. eCollection 2019 Jun. PMID 31158230
- [Derived] Merisaari H, Jambor I, Ettala O, Bostrom PJ, Montoya Perez I, Verho J, Kiviniemi A, Syvanen K, Kahkonen E, Eklund L, Pahikkala T, Vainio P, Saunavaara J, Aronen HJ, Taimen P. IMPROD biparametric MRI in men with a clinical suspicion of prostate cancer (IMPROD Trial): Sensitivity for prostate cancer detection in correlation with whole-mount prostatectomy sections and implications for focal therapy. J Magn Reson Imaging. 2019 Nov;50(5):1641-1650. doi: 10.1002/jmri.26727. Epub 2019 Mar 22. PMID 30903647